CLINICAL TRIAL: NCT05712551
Title: Diagnostic Agreement Among Expert Dermatopathologists on Skin Lesions Clinically Suspicious of Melanoma
Brief Title: Dermoscopy Augmented Histology Trial, Consensus Agreement Diagnosis Made by Dermatopathology Experts
Status: Enrolling by invitation | Type: Observational
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Louisa Bønløkke Nervil, Medical doctor, Herlev Hospital
Other Study IDs: AISC-DAHT, consensus agreement
Record Dates: First submitted 2023-01-16; First posted 2023-02-03 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Melanoma (Skin); Pigmented Lesions
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It has been suggested that pathologists' diagnostic accuracy and confidence could be improved if they gained access to additional clinical information and in-vivo clinical and dermoscopic images of melanocytic tumors. This study examines the effect of digital training for pathologists in interpreting dermoscopic and clinical skin tumor images. The primary outcome of the upcoming DAHT RCT (Dermoscopy Augmented Histology Trial, a randomized controlled trial) is the diagnostic value (accuracy, sensitivity, and specificity) for the intervention and control group. For this purpose, we need an expert agreeable MPATH-Dx classification and diagnosis for all DAHT cases. The DAHT consensus trial strives to establish this gold standard through a four-phased Delphi-like process.

Aim: To establish an expert agreeable MPTAH-Dx classification and diagnosis for all DAHT cases.

Data collection of DAHT cases: Department of plastic surgery, Herlev hospital, year 2020-2021

DAHT platform: Made in 2021-2023 by Melatech

Consensus agreement: Four dermatopathologists assess all DAHT cases, year 2023-2024

DETAILED DESCRIPTION:
Background Several publications suggest that the increasing melanoma incidence may partly be caused by histopathological overdiagnosis (Glasziou, 2020). Pathologists provide the current gold standard in skin lesion diagnostics (Elmore, 2017), most often primarily based on the interpretation of histological slides. Still, it has been suggested that pathologists' diagnostic accuracy and confidence could be improved if they gained access to additional clinical information and in-vivo clinical and dermoscopic images of melanocytic tumors (Scolyer, 2019) (Elder, 2018). This could help the pathologist generate a complete image of the lesion. However, interpreting clinical and dermoscopic images is challenging, and mastery typically requires several years of clinical experience (Ternov 2021). This learning journey can be significantly shortened if the trainee receives comprehensive training in pattern recognition for dermoscopy and clinical images, including immediate, accurate, and individualized feedback and access to a library with a large selection of skin lesion cases (Ericsson, 2015).

This study examines the effect of digital training for pathologists in interpreting dermoscopic and clinical skin tumor images.

Former studies have only focused on melanocytic lesions. Still, most pathologists will receive both melanocytic and pigmented non-melanocytic lesions (seborrheic keratoses, dermatofibromas, etc.) due to clinical suspicion of melanoma. This study includes an un-filtered selection of 211 clinically melanoma-suspect skin lesions excised at a specialized surgical department; this material is named the DAHT cases.

The primary outcome of the upcoming DAHT RCT (Dermoscopy Augmented Histology Trial, a randomized controlled trial) is the diagnostic value (accuracy, sensitivity, and specificity) for the intervention and control group. For this purpose, we need an MPATH-Dx classification and diagnosis for all DAHT cases agreed upon by experts in the field. The DAHT consensus agreement trial strives to establish this through a four-phased Delphi-like process.

Aim: To establish an expert agreeable MPTAH-Dx classification and diagnosis for all DAHT cases.

Method Case Database

Lesion data were collected from patients between 02.11.2020 and 22.01.2021 at the Department of Plastic Surgery, Herlev Hospital. Requirements for eligibility for the current study are:

The patient was referred through the clinical cancer pathways for melanoma. The lesion was excised upon evaluation by the plastic surgeon.

Patients received oral and written information about the project and were asked to sign a consent form before participation. The participation did not affect the included patients' treatment, diagnostics, or follow-up. Upon consent, the following information was collected for each lesion:

Clinical image Dermoscopic image Patient CPR-number (personal ID number) Sex and age of the patient Location of skin tumor (on a 3D avatar) Medical history (former treatment, congenital nevi, if pregnant, time of appearance of skin lesion, change in appearance, symptoms, former melanoma or other skin diseases, family history of melanoma, sun exposure within the last six months) After excision, the specimen was prepared for pathological examination and a representative hematoxylin-eosin stain, and, if available, a MelanA stain for each skin lesion was chosen for the study by an experienced dermatopathologist. These stains were subsequently digitized and coupled with the relevant information (dermoscopic and clinical image, tumor location, sex, age, lesion information, etc.). The CPR number was deleted, rendering the case anonymous. Each case is stored in a database under a random anonymous ID number.

Web-based IT platform

To maximize the number of pathologists included in the study, the investigators have developed an IT platform for the trial (The DAHT platform). The platform enables the following features:

Sign-in Automated randomization Login Case presentation Diagnosis of cases and subquestions Tracking The diagnostic options will be based on the standardized MPATH-Dx version 2.0 (Barnhill, 2023). After diagnosing the lesion, participating pathologists will rate both confidence and difficulty in the chosen diagnosis on a 6-step Likert scale. They will also be asked whether they want a second opinion and what tests/stains they need. The tracking feature will enable search pattern analysis, including time per diagnosis and percentage of time spent looking at histology stains, dermoscopic images, clinical images, and clinical information.

Consensus agreement The consensus agreement on the diagnosis of each case and MPATH-Dx classification will be reached through a Delphi-like process consisting of four phases. Four international well-acknowledged experts in dermatopathology have been invited to participate as the expert panel in this study.

Phase 1 - Online discussion When phase 1 has been concluded, all experts will be invited to an online discussion. Issues and suggestions regarding the DAHT cases and platform will be discussed during the meeting. The primary investigator will formulate a plan to remedy/accommodate these. If the expert group concludes that additional cases are required for the DAHT study, these will be collected by the primary investigator.

Phase 2 - Independent diagnostics All participating experts will be asked to independently review and diagnose all 211 DAHT cases. This will be facilitated through the DAHT platform (developed for the purpose), and the primary investigator will send regular reminders if needed. The website continuously saves the experts' progress, ensuring they can diagnose the 211 cases in small batches over 30 days. All experts will be asked to take notes regarding suggestions to improve the DAHT platform and DAHT dataset.

Phase 3 - Review of ambiguous cases An anonymous report with data from Phase 1 and a list of all ambiguous cases with less than 80% observer agreement and cases in which all experts are rated higher than four on difficulty and confidence will be emailed to the participating experts. The experts will be asked to reevaluate the ambiguous cases independently, with the data from phase 1 at hand. Similar to the previous phase, cases with less than 80% observer agreement/ a confidence and a difficulty level of four or more will go on to phase 4.

Phase 4 - Consensus discussion (online or physical) The primary investigator will facilitate a consensus agreement discussion among the experts regarding the most challenging cases where a disagreement persists beyond Phase 3. An anonymous report on data from Phase 3 will be available during this meeting.

ELIGIBILITY:
Inclusion Criteria:

* well-acknowledged expert in dermatopathology
* Invited by our group

Exclusion Criteria:

* Do not assess all DAHT cases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Experts in dermatopathology who are invited and willing to participate and, if necessary, discuss their diagnosis with other participants in an online meeting.r
Sampling Method: Non-Probability Sample
Enrollment: 4 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2024-12-29 (Estimated); Study Completion 2025-12-29 (Estimated)

PRIMARY OUTCOMES:
Gold standard diagnosis by using a Delphi-like process | 3 months
  Diagnostic agreement among participating experts in all DAHT cases with individual assessments and, later on, a discussion about ambiguous cases.

CONTACTS AND LOCATIONS:
Overall Officials: Lisbet Rosenkrantz Hôlmich, MD. prof., Study Director — Herlev University Hospital, Denmark
Locations (1):
- Herlev University Hospital, Herlev, Denmark

REFERENCES:
- [Background] Barnhill RL, Elder DE, Piepkorn MW, Knezevich SR, Reisch LM, Eguchi MM, Bastian BC, Blokx W, Bosenberg M, Busam KJ, Carr R, Cochran A, Cook MG, Duncan LM, Elenitsas R, de la Fouchardiere A, Gerami P, Johansson I, Ko J, Landman G, Lazar AJ, Lowe L, Massi D, Messina J, Mihic-Probst D, Parker DC, Schmidt B, Shea CR, Scolyer RA, Tetzlaff M, Xu X, Yeh I, Zembowicz A, Elmore JG. Revision of the Melanocytic Pathology Assessment Tool and Hierarchy for Diagnosis Classification Schema for Melanocytic Lesions: A Consensus Statement. JAMA Netw Open. 2023 Jan 3;6(1):e2250613. doi: 10.1001/jamanetworkopen.2022.50613. PMID 36630138
- [Result] Whiteman DC, Green AC, Olsen CM. The Growing Burden of Invasive Melanoma: Projections of Incidence Rates and Numbers of New Cases in Six Susceptible Populations through 2031. J Invest Dermatol. 2016 Jun;136(6):1161-1171. doi: 10.1016/j.jid.2016.01.035. Epub 2016 Feb 20. PMID 26902923
- [Result] Glasziou PP, Jones MA, Pathirana T, Barratt AL, Bell KJ. Estimating the magnitude of cancer overdiagnosis in Australia. Med J Aust. 2020 Mar;212(4):163-168. doi: 10.5694/mja2.50455. Epub 2019 Dec 19. PMID 31858624
- [Result] Elmore JG, Barnhill RL, Elder DE, Longton GM, Pepe MS, Reisch LM, Carney PA, Titus LJ, Nelson HD, Onega T, Tosteson ANA, Weinstock MA, Knezevich SR, Piepkorn MW. Pathologists' diagnosis of invasive melanoma and melanocytic proliferations: observer accuracy and reproducibility study. BMJ. 2017 Jun 28;357:j2813. doi: 10.1136/bmj.j2813. PMID 28659278
- [Result] Scolyer RA, Soyer HP, Kelly JW, James C, McLean CA, Coventry BJ, Ferguson PM, Rawson RV, Mar VJ, de Menezes SL, Fishburn P, Stretch JR, Lee S, Thompson JF. Improving diagnostic accuracy for suspicious melanocytic skin lesions: New Australian melanoma clinical practice guidelines stress the importance of clinician/pathologist communication. Aust J Gen Pract. 2019 Jun;48(6):357-362. doi: 10.31128/AJGP-11-18-4759. PMID 31220881
- [Result] Ferrara G, Argenyi Z, Argenziano G, Cerio R, Cerroni L, Di Blasi A, Feudale EA, Giorgio CM, Massone C, Nappi O, Tomasini C, Urso C, Zalaudek I, Kittler H, Soyer HP. The influence of clinical information in the histopathologic diagnosis of melanocytic skin neoplasms. PLoS One. 2009;4(4):e5375. doi: 10.1371/journal.pone.0005375. Epub 2009 Apr 30. PMID 19404399
- [Result] Bedlow AJ, Cliff S, Melia J, Moss SM, Seyan R, Harland CC. Impact of skin cancer education on general practitioners' diagnostic skills. Clin Exp Dermatol. 2000 Mar;25(2):115-8. doi: 10.1046/j.1365-2230.2000.00590.x. PMID 10733633
- [Result] Badertscher N, Tandjung R, Senn O, Kofmehl R, Held U, Rosemann T, Hofbauer GF, Wensing M, Rossi PO, Braun RP. A multifaceted intervention: no increase in general practitioners' competence to diagnose skin cancer (minSKIN) - randomized controlled trial. J Eur Acad Dermatol Venereol. 2015 Aug;29(8):1493-9. doi: 10.1111/jdv.12886. Epub 2014 Dec 10. PMID 25491768
- [Result] Ternov NK, Vestergaard T, Holmich LR, Karmisholt K, Wagenblast AL, Klyver H, Hald M, Schollhammer L, Konge L, Chakera AH. Reliable test of clinicians' mastery in skin cancer diagnostics. Arch Dermatol Res. 2021 May;313(4):235-243. doi: 10.1007/s00403-020-02097-8. Epub 2020 Jun 28. PMID 32596742